CLINICAL TRIAL: NCT06486675
Title: The Effect of Face-to-Face Breastfeeding Counseling Training on Breast Milk Perception
Brief Title: Breastfeeding Counseling Training on Breast Milk Perception and Baby Feeding Attitudes
Acronym: EFFBCTBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, PhD, Assist. Prof. Dr, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIU3
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: MİDWİFERY STUDENT
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education (Experimental): The pre-test data from the students in the experimental group were collected in the first lesson via the Google form created using the "Personal Introduction Form", "Adults' Perception Scale on Breast Milk (ASAÖ)" and "Iowa Infant Nutrition Attitude Scale (IOWA)", and the first and The second will be sent to the students by the authors. The first question was asked, "Are you willing to participate in this research?" Those who say yes will read and fill out this form themselves. At the end of the 14-week course period, post-test data will be obtained using the same method.
  Interventions: Other: education
- control group (No Intervention): 640 / 5.000 The pre-test data from the students in the control group is a survey form created by the third author using the "Personal Introduction Form", "Adults' Perception Scale on Mother's Milk (ASAÖ)" and "Infant Nutrition Attitude Scale (IOWA)" before a suitable lesson in the first week of the semester. The form link will be created and sent to the students by the third author via WhatsApp messaging application. The first question was asked, "Are you willing to participate in this research?" Those who say yes will read and fill out this form themselves. At the end of the 14-week course period, the post-test data will be obtained by the third author using the same method.

INTERVENTIONS:
Other: education — breastfeeding consultant training
  Other Names: other
  Arms: education

SUMMARY:
This research will be conducted to determine the effect of face-to-face breastfeeding counseling training on breast milk perception and infant nutrition attitudes.The population of this semi-experimental research consisted of students who took the Breastfeeding Consultancy course at Kahramanmaraş Sütçü İmam University Faculty of Health Sciences (n=49) and 3rd year students who did not take this course at İnönü University Faculty of Health Sciences (n=47). "Personal Introduction Form", "Adults' Perception Scale on Breast Milk (ASAÖ)" and "Infant Nutrition Attitude Scale (IOWA)" will be used to collect pre-test and post-test data. Pretest data were obtained in the first lesson of the semester in both groups. Participants in the experimental group were given training consisting of breastfeeding counseling course content for 14 weeks. The control group was not given any training on this subject. At the end of the semester, post-test measurements will be made to both groups simultaneously and with the same measurement tools.

DETAILED DESCRIPTION:
The rich nutrients contained in breast milk ensure the survival and healthy growth of the newborn . Apart from being a nutrient for the mother and the newborn, breast milk and breastfeeding have many benefits in terms of psychological, social development, immune system, developmental, spiritual, social and financial benefits . It is recommended that the baby should not be breastfed without additional food for the first 6 months . However, although the rate of breastfeeding in Turkey is 98%, the rate of babies being fed only breast milk for the first 6 months is reported to be 41% in the Turkey Population and Health Survey (TDHS)-2018 report. It is very important that breastfeeding begins and continues successfully. However, the breastfeeding process can be affected by many factors related to mother and baby. The mother may not be able to cope alone with some challenging factors such as breast rejection, frequent crying, dissatisfaction after breastfeeding, small amounts of defecation, and insufficient breast milk. In case of possible or real problems with breastfeeding, breastfeeding counseling is required . Providing breastfeeding education and counseling is one of the most important roles and responsibilities of midwives during pregnancy, birth and postpartum . The breastfeeding support that the mother receives from midwives greatly affects breastfeeding decisions. Effective breastfeeding support increases breastfeeding duration and success . Midwifery students are given training on breast milk and breastfeeding in accordance with the Midwifery National Core Education Program (EUÇEP). The purpose of breastfeeding counseling training is to train people to evaluate and manage breastfeeding problems . During the breastfeeding consultancy process; The aim is to support mothers in breastfeeding, to reveal the causes of breast milk insufficiency and to implement practices to increase breast milk However, it has been emphasized in the literature that midwives' breastfeeding counseling is not at the desired level . Breastfeeding counseling course is not included in the curriculum of midwifery departments of every university in Turkey . Studies have also shown that mothers are not always satisfied with the breastfeeding support they receive from midwives after birth A quality education based on evidence-based breastfeeding counseling is required for midwives and midwifery students to provide effective breastfeeding support to breastfeeding women tfeeding is effective in successfully maintaining the self-efficacy and breastfeeding behavior of mothers during the lactation process . It is thought that with this research, the curriculum of the midwifery department of the breastfeeding counseling course will be reviewed and will contribute positively to the increase in breastfeeding rates in our country in the future. The purpose of this research is to determine the effect of breastfeeding counseling training on midwifery students' perception of breast milk and infant feeding attitudes.

ELIGIBILITY:
Inclusion Criteria:

* being a midwifery student no communication problems Healthy Volunteers

Exclusion Criteria:

* communication problems

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
First Measurement: 1.602 / 5.000 First Measurement:Adult Perception Scale on Breast Milk | 3 MONTH
  Adults' Perception Scale on Breast Milk is a five-point Likert-type, one-dimensional scale consisting of 30 items. The minimum total score to be obtained from the scale is 30 and the maximum is 150 points. As adults' ASAS score increases, it shows that their perception of breast milk is at a good level. C
Second Measurement:Baby Nutrition Attitude Scale (IOWA) | 3 month
  Baby Nutrition Attitude Scale is a scale created by De La Moraave Russell (1999) to predict participants' attitudes towards breastfeeding and the duration of breastfeeding (De La Mora,2019). The scale consists of 17 items and is a 5-point Likert type scale. 8 items in the scale are about formula feeding, and 9 items are about breastfeeding. Scoring of items related to formula nutrition is done by reverse scoring. The total score to be received varies between 17 and 85, and a low score indicates that the participant has a positive attitude towards bottle feeding, and a high score indicates that the participant has a positive attitude towards breastfeeding.

IPD SHARING:
Plan to Share IPD: No